CLINICAL TRIAL: NCT01287520
Title: Phase 1 Dose Escalation Study of LY2090314 in Patients With Advanced or Metastatic Cancer in Combination With Pemetrexed and Carboplatin
Brief Title: A Study of LY2090314 in Patients With Advanced or Metastatic Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 11613; I2H-MC-JWYA (Other: Eli Lilly and Company)
Record Dates: First submitted 2011-01-28; First posted 2011-02-01 (Estimated); Results first posted 2019-02-25 (Actual); Last update posted 2019-02-25 (Actual); Status verified 2018-10

CONDITIONS: Advanced Cancer
MeSH Terms: interventions — 3-(9-fluoro-2-(piperidin-1-ylcarbonyl)-1,2,3,4-tetrahydro(1,4)diazepino(6,7,1-hi)indol-7-yl)-4-imidazo(1,2-a)pyridin-3-yl-1H-pyrrole-2,5-dione; Pemetrexed; Carboplatin; Ranitidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- LY2090314/pemetrexed/carboplatin (Experimental): Part A, Cycle 1 (28 days): Intravenous doses of LY2090314 starting at 10 milligram (mg) were given on Day 1 followed by 10 mg LY2090314, 500 milligram per square meter (mg/m^2) pemetrexed (intravenous dose), and 5 or 6 area under the concentration-time curve (AUC) intravenous dose of carboplatin on Day 8.
  Part A, Cycle 2 (21 days): Pemetrexed and carboplatin given on Day 1 at the same dose administered in Cycle 1.
  Part A, Cycle 3 (21 days) and beyond: LY2090314, Pemetrexed and carboplatin were given on Day 1 at the same dose administered in Cycle 1. LY2090314 doses were escalated until the maximum tolerated dose (MTD) was reached.
  Part B: Dose determined in Part A was administered. Participants were allowed to continue the combination treatment if they were receiving therapeutic benefit until they fulfilled one of the criteria for discontinuation.
  Interventions: Drug: LY2090314; Drug: pemetrexed; Drug: Carboplatin; Other: ranitidine

INTERVENTIONS:
Drug: LY2090314 — Administered intravenously
Drug: pemetrexed — Administered intravenously
  Other Names: Alimta; LY231514
Drug: Carboplatin — Administered intravenously
Other: ranitidine — Per I2H-MC-JWYA Protocol Amendment (d) approved 11 March 2010, 50 mg ranitidine given as pretreatment to LY2090314 for stomach pain.

SUMMARY:
The purpose of this study is to determine a recommended Phase 2 dose and dosing regimen of LY2090314 in combination with pemetrexed and carboplatin in patients with advanced/metastatic cancer. Part A of this study will consist of dose escalation of the study regimen, and Part B will consist of an expanded cohort to confirm the dose provided from Part A.

ELIGIBILITY:
Inclusion Criteria:

* Have a performance status of less than or equal to 2 on the Eastern Cooperative Oncology Group (ECOG) scale
* Have a life expectancy of greater than or equal to 12 weeks
* Males and females with reproductive potential agree to use medically approved contraceptive precautions during the trial and for 3 months following the last dose of study drug
* Have histological or cytological evidence of a diagnosis of cancer that is advanced and/or metastatic disease for which no proven effective therapy exists
* Have the presence of measurable or nonmeasurable disease as defined by the Response Evaluation Criteria in Solid Tumors (RECIST)
* Have adequate hematologic, hepatic, and renal function
* Have discontinued all previous therapies for cancer, including chemotherapy, radiotherapy, cancer-related hormonal therapy, or other investigational therapy for at least 30 days (6 weeks for mitomycin-C or nitrosoureas) prior to study enrollment and recovered from the acute effects of therapy.

Exclusion Criteria:

* Have received treatment within 30 days of the initial dose of study drug with a drug that has not received regulatory approval for any indication
* Have serious preexisting medical conditions (left to discretion of investigator)
* Have one of the following conduction abnormalities: Corrected time between start of Q wave and end of T wave (QTc) prolongation >450 millisecond (msec) on screening electrocardiogram (ECG), previous history of QTc prolongation with another medication that required discontinuation, congenital long-QT-syndrome, or left bundle branch block (LBBB)
* Are taking any concomitant medication that may cause QTc prolongation, or induce Torsades de Pointes
* Have systolic blood pressure greater than or equal to 140 millimeters of Mercury (mm Hg), and diastolic blood pressure greater than or equal to 90 mm Hg that is not controlled by medical therapy
* Have serious cardiac condition, such as myocardial infarction within 6 months, angina, or heart disease, as defined by the New York Heart Association Class II or higher; have history of arrhythmia that is symptomatic or requires treatment
* Have chronic atrial fibrillation and/or bradycardia
* Have uncorrected electrolyte disorders including potassium <3.4 molar equivalent per liter (mEq/L) (<3.4 millimole per liter [mmol/l]), calcium <8.4 milligram per deciliter (mg/dL) (2.1 mmol/L), or magnesium <1.2 mg/dL (<0.62 mmol/L)
* Have symptomatic central nervous system (CNS) malignancy or metastasis (screening not required)
* Have a hematologic malignancy
* Females who are pregnant or lactating

Min Age: 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2007-11; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (2):
- United States (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tampa, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nashville, Tennessee

REFERENCES:
- [Derived] Gray JE, Infante JR, Brail LH, Simon GR, Cooksey JF, Jones SF, Farrington DL, Yeo A, Jackson KA, Chow KH, Zamek-Gliszczynski MJ, Burris HA 3rd. A first-in-human phase I dose-escalation, pharmacokinetic, and pharmacodynamic evaluation of intravenous LY2090314, a glycogen synthase kinase 3 inhibitor, administered in combination with pemetrexed and carboplatin. Invest New Drugs. 2015 Dec;33(6):1187-96. doi: 10.1007/s10637-015-0278-7. Epub 2015 Sep 25. PMID 26403509

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The reasons for discontinuation listed in the participant flow are the reasons the participant discontinued treatment and a participant was considered to have "completed" the trial if they discontinued treatment due to progressive disease or an adverse event.
Groups:
- LY 10/Carb 5/Pem 500 (Cohort 1): * Cycle 1 Day 1 of 28-day cycle: 10 milligrams (mg) LY2090314 (LY) administered by intravenous infusion.
  * Cycle 1 Day 8 of 28-day cycle: 500 milligrams per meter squared (mg/m^2) pemetrexed (Pem) administered by intravenous infusion followed by Area Under the Time Curve (AUC) 5 milligrams per milliliter times minutes (mg/mL * min) carboplatin (Carb) administered by intravenous infusion.
  * Cycle 2 and beyond: Day 1 of 21-day cycle: 500 mg/m^2 Pem administered by intravenous infusion followed by AUC 5 mg/mL * min Carb administered by intravenous infusion followed by 10 mg LY2090314 administered by intravenous infusion.
- LY 10/Carb 6/Pem 500 (Cohort 2): * Cycle 1 Day 1 of 28-day cycle: 10 mg LY2090314 by intravenous infusion.
  * Cycle 1 Day 8 of 28-day cycle: 500 mg/m^2 Pem by intravenous infusion followed by AUC 6 mg/mL * min Carb by intravenous infusion.
  * Cycle 2 and beyond: Day 1 of 21-day cycle: 500 mg/m^2 Pem by intravenous infusion followed by AUC 6 mg/mL * min Carb by intravenous infusion followed by 10 mg LY2090314 by intravenous infusion.
- LY 20/Carb 6/Pem 500 (Cohort 3): * Cycle 1 Day 1 of 28-day cycle: 20 mg LY2090314 by intravenous infusion.
  * Cycle 1 Day 8 of 28-day cycle: 500 mg/m^2 Pem by intravenous infusion followed by AUC 6 mg/mL * min Carb by intravenous infusion.
  * Cycle 2 and beyond: Day 1 of 21-day cycle: 500 mg/m^2 Pem by intravenous infusion followed by AUC 6 mg/mL * min Carb by intravenous infusion followed by 20 mg LY2090314 by intravenous infusion.
- LY 40/Carb 6/Pem 500 (Cohort 4): * Cycle 1 Day 1 of 28-day cycle: 40 mg LY2090314 by intravenous infusion.
  * Cycle 1 Day 8 of 28-day cycle 500 mg/m^2 Pem by intravenous infusion followed by AUC 6 mg/mL * min Carb by intravenous infusion followed by 40 mg LY2090314 by intravenous infusion.
  * Cycle 2 Day 1 of 21-day cycle: AUC 6 mg/mL * min Carb by intravenous infusion followed by 500 mg/m^2 Pem by intravenous infusion.
  * Cycle 3 and beyond: Day 1 of 21 day cycle: 500 mg/m^2 Pem by intravenous infusion followed by AUC 6 mg/mL * min Carb by intravenous infusion followed by 40 mg LY2090314 by intravenous infusion.
- LY 80/Carb 6/Pem 500 (Cohort 5): * Cycle 1 Day 1 of 28 -ay cycle: 80 mg LY2090314 by intravenous infusion.
  * Cycle 1 Day 8 of 28-day cycle 500 mg/m^2 Pem by intravenous infusion followed by AUC 6 mg/mL * min Carb by intravenous infusion followed by 80 mg LY2090314 by intravenous infusion.
  * Cycle 2 Day 1 of 21-day cycle: AUC 6 mg/mL * min Carb by intravenous infusion followed by 500 mg/m^2 Pem by intravenous infusion.
  * Cycle 3 up and beyond: Day 1 of 21 day cycle: 500 mg/m^2 Pem by intravenous infusion followed by AUC 6 mg/mL * min Carb by intravenous infusion followed by 80 mg LY2090314 by intravenous infusion
- LY 120/Carb 6/Pem 500 -(Cohort 6): * Cycle 1 Day 1 of 28-day cycle: 120 mg LY2090314 by intravenous infusion.
  * Cycle 1 Day 8 of 28-day cycle 500 mg/m^2 Pem by intravenous infusion followed by AUC 6 mg/mL * min Carb by intravenous infusion followed by 120 mg LY2090314 by intravenous infusion.
  * Cycle 2 Day 1 of 21-day cycle: AUC 6 mg/mL * min Carb by intravenous infusion followed by 500 mg/m^2 Pem by intravenous infusion.
  * Cycle 3 and beyond: Day 1 of 21-day cycle: 500 mg/m^2 Pem by intravenous infusion followed by AUC 6 mg/mL * min Carb by intravenous infusion followed by 120 mg LY2090314 by intravenous infusion.
- LY 80/Carb 6/Pem 500 + R50 (Cohort 7): * Cycle 1 Day 1 of 28-day cycle: pretreated with 50 mg ranitidine (R50) intravenous, 80 mg LY2090314 by intravenous infusion.
  * Cycle 1 Day 8 of 28-day cycle 500 mg/m^2 Pem by intravenous infusion followed by AUC 6 mg/mL * min Carb intravenous infusion followed by 50 mg ranitidine intravenous pretreatment and 80 mg LY2090314 by intravenous infusion.
  * Cycle 2 Day 1 of 21-day cycle: AUC 6 mg/mL * min Carb by intravenous infusion followed by 500 mg/m^2 Pem IV infusion.
  * Cycle 3 and beyond: Day 1 of 21-day cycle: 500 mg/m^2 Pem by intravenous infusion followed by AUC 6 mg/mL * min Carb by intravenous infusion followed by 50 mg ranitidine intravenous pretreatment and 80 mg LY2090314 intravenous infusion.
  Based on I2H-MC-JWYA Protocol Amendment (d) approved 11 March 2010, 50 mg ranitidine was given as a pretreatment to LY2090314 as prophylaxis for stomach pain.
- LY 60/Carb 6/Pem 500 + R50 (Cohort 8): * Cycle 1 Day 1 of 28-day cycle: pretreated with 50 mg ranitidine intravenous, 60 mg LY2090314 by IV infusion.
  * Cycle 1 Day 8 of 28-day cycle 500 mg/m^2 Pem by intravenous infusion followed by AUC 6mg/mL * min Carb intravenous infusion followed by 50 mg ranitidine intravenous pretreatment and 60 mg LY2090314 by intravenous infusion.
  * Cycle 2 Day 1 of 21-day cycle: AUC 6 mg/mL * min Carb by intravenous infusion followed by 500 mg/m^2 Pem intravenous infusion.
  * Cycle 3 and beyond: Day 1 of 21-day cycle: 500 mg/m^2 Pem by intravenous infusion followed by AUC 6 mg/mL * min Carb by intravenous infusion followed by 50 mg ranitidine intravenous pretreatment and 60 mg LY2090314 intravenous infusion.
  Based on I2H-MC-JWYA Protocol Amendment (d) approved 11 March 2010, 50 mg ranitidine was given as a pretreatment to LY2090314 as prophylaxis for stomach pain.
- LY 40/Carb 6/Pem 500 + R50 (Cohort 9): * Cycle 1 Day 1 of 28-day cycle: pretreated with 50 mg ranitidine intravenous, 40 mg LY2090314 by intravenous infusion.
  * Cycle 1 Day 8 of 28-day cycle 500 mg/m^2 Pem by intravenous infusion followed by AUC 6 mg/mL * min Carb intravenous infusion followed by 50 mg ranitidine intravenous pretreatment and 40 mg LY2090314 by intravenous infusion.
  * Cycle 2 Day 1 of 21-day cycle: AUC 6 mg/mL * min Carb by intravenous infusion followed by 500 mg/m^2 Pem intravenous infusion.
  * Cycle 3 and beyond: Day 1 of 21-day cycle: 500 mg/m^2 Pem by intravenous infusion followed by AUC 6 mg/mL * min Carb by intravenous infusion followed by 50 mg ranitidine IV pretreatment and 40 mg LY2090314 intravenous infusion.
  Based on I2H-MC-JWYA Protocol Amendment (d) approved 11 March 2010, 50 mg ranitidine was given as a pretreatment to LY2090314 as prophylaxis for stomach pain.
Period: Overall Study
Arm/Group | LY 10/Carb 5/Pem 500 (Cohort 1) | LY 10/Carb 6/Pem 500 (Cohort 2) | LY 20/Carb 6/Pem 500 (Cohort 3) | LY 40/Carb 6/Pem 500 (Cohort 4) | LY 80/Carb 6/Pem 500 (Cohort 5) | LY 120/Carb 6/Pem 500 -(Cohort 6) | LY 80/Carb 6/Pem 500 + R50 (Cohort 7) | LY 60/Carb 6/Pem 500 + R50 (Cohort 8) | LY 40/Carb 6/Pem 500 + R50 (Cohort 9)
Started | 3 | 7 (One participant who received study drug but did not complete Cycle 1 was replaced.) | 5 | 7 (One participant who received study drug but did not complete Cycle 1 was replaced.) | 3 | 4 | 2 | 5 | 5
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 3 | 7 | 5 | 7 | 3 | 4 | 2 | 5 | 5
Not completed — Adverse Event | 2 | 2 | 2 | 1 | 1 | 2 | 0 | 2 | 0
Not completed — Physician Decision | 1 | 1 | 2 | 0 | 1 | 1 | 0 | 1 | 0
Not completed — Progressive disease | 0 | 4 | 1 | 6 | 1 | 0 | 2 | 2 | 4
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: All randomized participants who received at least 1 dose of study drug.
Groups:
- LY 10/Carb 5/Pem 500 (Cohort 1): * Cycle 1 Day 1 of 28-day cycle: 10 mg LY2090314 by intravenous infusion.
  * Cycle 1 Day 8 of 28-day cycle: 500 mg/m^2 Pem by intravenous infusion followed by AUC 5 mg/mL * min Carb by intravenous infusion.
  * Cycle 2 up to Cycle 9: Day 1 of 21-day cycle: 500 mg/m^2 Pem by intravenous infusion followed by AUC 5 mg/mL * min Carb by intravenous infusion followed by 10 mg LY2090314 by intravenous infusion.
- LY 10/Carb 6/Pem 500 (Cohort 2): * Cycle 1 Day 1 of 28-day cycle: 10 mg LY2090314 by intravenous infusion.
  * Cycle 1 Day 8 of 28-day cycle: 500 mg/m^2 Pem by intravenous infusion followed by AUC 6 mg/mL * min Carb by intravenous infusion.
  * Cycle 2 up to Cycle 9: Day 1 of 21-day cycle: 500 mg/m^2 Pem by intravenous infusion followed by AUC 6 mg/mL * min Carb by intravenous infusion followed by 10 mg LY2090314 by intravenous infusion.
- LY 20/Carb 6/Pem 500 (Cohort 3): * Cycle 1 Day 1 of 28-day cycle: 20 mg LY2090314 by intravenous infusion.
  * Cycle 1 Day 8 of 28-day cycle: 500 mg/m^2 Pem by intravenous infusion followed by AUC 6 mg/mL * min Carb by intravenous infusion.
  * Cycle 2 up to Cycle 9: Day 1 of 21-day cycle: 500 mg/m^2 Pem by intravenous infusion followed by AUC 6 mg/mL * min Carb by intravenous infusion followed by 20 mg LY2090314 by intravenous infusion.
- LY 40/Carb 6/Pem 500 (Cohort 4): * Cycle 1 Day 1 of 28-day cycle: 40 mg LY2090314 by intravenous infusion.
  * Cycle 1 Day 8 of 28-day cycle 500 mg/m^2 Pem by intravenous infusion followed by AUC 6 mg/mL * min Carb by intravenous infusion followed by 40 mg LY2090314 by intravenous infusion.
  * Cycle 2 Day 1 of 21-day cycle: AUC 6 mg/mL * min Carb by intravenous infusion followed by 500 mg/m^2 Pem by intravenous infusion.
  * Cycle 3 up to Cycle 9: Day 1 of 21-day cycle: 500 mg/m^2 Pem by intravenous infusion followed by AUC 6 mg/mL * min Carb by intravenous infusion followed by 40 mg LY2090314 by intravenous infusion.
- LY 80/Carb 6/Pem 500 (Cohort 5): * Cycle 1 Day 1 of 28-day cycle: 80 mg LY2090314 by intravenous infusion.
  * Cycle 1 Day 8 of 28-day cycle 500 mg/m^2 Pem by intravenous infusion followed by AUC 6 mg/mL * min Carb by intravenous infusion followed by 80 mg LY2090314 by intravenous infusion.
  * Cycle 2 Day 1 of 21-day cycle: AUC 6 mg/mL * min Carb by intravenous infusion followed by 500 mg/m^2 Pem by intravenous infusion.
  * Cycle 3 up to Cycle 9: Day 1 of 21-day cycle: 500 mg/m^2 Pem by intravenous infusion followed by AUC 6 mg/mL * min Carb by intravenous infusion followed by 80 mg LY2090314 by intravenous infusion.
- LY 120/Carb 6/Pem 500 (Cohort 6): * Cycle 1 Day 1 of 28-day cycle: 120 mg LY2090314 by intravenous infusion.
  * Cycle 1 Day 8 of 28-day cycle 500 mg/m^2 Pem by intravenous infusion followed by AUC 6 mg/mL * min Carb by intravenous infusion followed by 120 mg LY2090314 by intravenous infusion.
  * Cycle 2 Day 1 of 21-day cycle: AUC 6 mg/mL * min Carb by intravenous infusion followed by 500 mg/m^2 Pem by intravenous infusion.
  * Cycle 3 up to Cycle 9: Day 1 of 21-day cycle: 500 mg/m^2 Pem by intravenous infusion followed by AUC 6 mg/mL * min Carb by intravenous infusion followed by 120 mg LY2090314 by intravenous infusion.
- LY 80/Carb 6/Pem 500 + R50 (Cohort 7): * Cycle 1 Day 1 of 28-day cycle: pretreated with 50 mg ranitidine intravenous, 80 mg LY2090314 by intravenous infusion.
  * Cycle 1 Day 8 of 28-day cycle 500 mg/m^2 Pem by intravenous infusion followed by AUC 6mg/mL * min Carb intravenous infusion followed by 50 mg ranitidine intravenous pretreatment and 80 mg LY2090314 by intravenous infusion.
  * Cycle 2 Day 1 of 21-day cycle: AUC 6 mg/mL * min Carb by intravenous infusion followed by 500 mg/m^2 Pem intravenous infusion.
  * Cycle 3 up to Cycle 10: Day 1 of 21-day cycle: 500 mg/m^2 Pem by intravenous infusion followed by AUC 6 mg/mL * min Carb by intravenous infusion followed by 50 mg ranitidine intravenous pretreatment and 80 mg LY2090314 intravenous infusion.
  Based on I2H-MC-JWYA Protocol Amendment (d) approved 11 March 2010, 50 mg ranitidine was given as a pretreatment to LY2090314 as prophylaxis for stomach pain.
- LY 60/Carb 6/Pem 500 + R50 (Cohort 8): * Cycle 1 Day 1 of 28-day cycle: pretreated with 50 mg ranitidine intravenous, 60 mg LY2090314 by intravenous infusion.
  * Cycle 1 Day 8 of 28-day cycle 500 mg/m^2 Pem by intravenous infusion followed by AUC 6mg/mL * min Carb intravenous infusion followed by 50 mg ranitidine intravenous pretreatment and 60 mg LY2090314 by intravenous infusion.
  * Cycle 2 Day 1 of 21-day cycle: AUC 6 mg/mL * min Carb by intravenous infusion followed by 500 mg/m^2 Pem intravenous infusion.
  * Cycle 3 up to Cycle 9: Day 1 of 21-day cycle: 500 mg/m^2 Pem by intravenous infusion followed by AUC 6 mg/mL * min Carb by intravenous infusion followed by 50 mg ranitidine intravenous pretreatment and 60 mg LY2090314 intravenous infusion.
  Based on I2H-MC-JWYA Protocol Amendment (d) approved 11 March 2010, 50 mg ranitidine was given as a pretreatment to LY2090314 as prophylaxis for stomach pain.
- LY 40/Carb 6/Pem 500 + R50 (Cohort 9): * Cycle 1 Day 1 of 28-day cycle: pretreated with 50 mg ranitidine intravenous, 40 mg LY2090314 by intravenous infusion.
  * Cycle 1 Day 8 of 28-day cycle 500 mg/m^2 Pem by intravenous infusion followed by AUC 6mg/mL * min Carb intravenous infusion followed by 50 mg ranitidine intravenous pretreatment and 40 mg LY2090314 by intravenous infusion.
  * Cycle 2 Day 1 of 21-day cycle: AUC 6 mg/mL * min Carb by intravenous infusion followed by 500 mg/m^2 Pem intravenous infusion.
  * Cycle 3 up to Cycle 9: Day 1 of 21-day cycle: 500 mg/m^2 Pem by intravenous infusion followed by AUC 6 mg/mL * min Carb by intravenous infusion followed by 50 mg ranitidine intravenous pretreatment and 40 mg LY2090314 intravenous infusion.
  Based on I2H-MC-JWYA Protocol Amendment (d) approved 11 March 2010, 50 mg ranitidine was given as a pretreatment to LY2090314 as prophylaxis for stomach pain.
- Total: Total of all reporting groups
Arm/Group | LY 10/Carb 5/Pem 500 (Cohort 1) | LY 10/Carb 6/Pem 500 (Cohort 2) | LY 20/Carb 6/Pem 500 (Cohort 3) | LY 40/Carb 6/Pem 500 (Cohort 4) | LY 80/Carb 6/Pem 500 (Cohort 5) | LY 120/Carb 6/Pem 500 (Cohort 6) | LY 80/Carb 6/Pem 500 + R50 (Cohort 7) | LY 60/Carb 6/Pem 500 + R50 (Cohort 8) | LY 40/Carb 6/Pem 500 + R50 (Cohort 9) | Total
Number analyzed (Participants) | 3 | 7 | 5 | 7 | 3 | 4 | 2 | 5 | 5 | 41
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.81 (11.88) | 55.27 (9.19) | 59.31 (5.62) | 58.32 (8.95) | 57.35 (7.59) | 56.73 (7.52) | 55.39 (9.86) | 58.78 (9.06) | 61.35 (4.41) | 57.79 (7.65)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 5 | 3 | 2 | 0 | 0 | 3 | 0 | 18
  Male | 1 | 4 | 0 | 4 | 1 | 4 | 2 | 2 | 5 | 23
Race/Ethnicity, Customized [Number; unit: participants]
  African | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 2
  Caucasian | 3 | 6 | 4 | 7 | 2 | 4 | 2 | 5 | 5 | 38
  Hispanic | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 3 | 7 | 5 | 7 | 3 | 4 | 2 | 5 | 5 | 41
Body Surface Area [Mean (Standard Deviation); unit: meters squared (m^2)] | 1.76 (0.11) | 2.10 (0.13) | 1.66 (0.14) | 1.94 (0.29) | 1.77 (0.46) | 2.11 (0.33) | 2.07 (0.14) | 1.90 (0.30) | 2.04 (0.15) | 1.94 (0.27)
Eastern Cooperative Oncology Group (ECOG) performance [Number; unit: participants] — ECOG - Classified participants according to their functional impairment. Scores ranged from 0 to 5: 0=Fully Active, No Restrictions; 1=Ambulatory, Able to Perform Light Work Activities (for example, light house work), Restricted Strenuous Activity; 2=Ambulatory, All Self Care, No Work Activities; 3=Partially Confined to Bed (>50% of waking hours), Limited Self Care; 4=Completely Disabled, Totally Bedridden; 5=Death
  participants
    0 | 3 | 5 | 5 | 7 | 2 | 4 | 2 | 3 | 5 | 36
    1 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 5
Basis of Diagnosis [Number; unit: participants]
  Cytological | 1 | 1 | 1 | 1 | 2 | 0 | 1 | 1 | 0 | 8
  Histopathological | 2 | 6 | 4 | 6 | 1 | 4 | 1 | 4 | 5 | 33
Initial Pathological Tumor Diagnosis [Number; unit: participants]
  Mesothelioma | 2 | 3 | 1 | 0 | 0 | 1 | 0 | 1 | 1 | 9
  Non-small cell lung carcinoma (NSCLC) | 0 | 0 | 3 | 1 | 1 | 0 | 0 | 1 | 1 | 7
  Leimyosarcoma | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 3
  Esophagus | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 3
  Lung adenocarcinoma | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 3
  Rectum | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2
  Small cell lung carcinoma (SCLC) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 2
  Gastric | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 2
  Head and neck | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Adenocarcinoma not otherwise specified (NOS) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Colon | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Breast | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
  Pancreas | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
  Cancer NOS | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
  Gall bladder | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
  Thymoma | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
  Adenoid | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
  Bile duct | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Recommended LY2090314 Dose for Phase 2 Studies (Maximum Tolerated Dose [MTD])
Description: Recommended Phase 2 MTD was determined, when a dose limiting toxicity (DLT) occurred in 1 of 3 participants, the cohort was to be expanded to 6 participants. If a DLT occurred in 2 or more participants, accrual to the cohort was stopped, as the MTD was exceeded. A DLT was defined as an adverse event (AE) occurring in Cycle 1 (28 days) that was possibly related to study drug and met 1 of the following criteria: According to the National Cancer Institute's (NCI) Common Terminology Criteria for Adverse Events (CTCAE) v3.0, ≥Grade 3 nonhematologic toxicity (except for nausea/vomiting without maximal symptomatic/prophylactic treatment) possibly or likely related to the study medication;CTCAE Grade 4 hematological toxicity of >5 days duration; Febrile neutropenia; CTCAE Grade 4 thrombocytopenia; CTCAE ≥Grade 2 thrombocytopenia plus bleeding; CTCAE ≥Grade 3 prolonged QTc interval.
Time Frame: Baseline up to Day 28 (Cycle 1)
Population: Safety population: all participants who have received at least 1 dose of the study drug.
Measure: Number; unit: milligrams (mg)
Groups:
- LY2090314/Pemetrexed/Carboplatin: Cycle 1 (28 days)
  Cohorts 1 to 3
  * Cycle 1 Day 1: 10-20 mg LY2090314 by intravenous infusion.
  * Cycle 1 Day 8: 500 mg/m^2 Pem by intravenous infusion followed by AUC 5 or 6 mg/mL * min Carb by intravenous infusion.
  Cohorts 4 to 9, Cohorts 7 to 9 were pretreated with 50 mg ranitidine intravenous-Cycle 1 Day 1: 40-120 mg LY2090314 by intravenous infusion.
  -Cycle 1 Day 8: 500 mg/m^2 by Pem intravenous infusion followed by AUC 6 mg/mL * min Carb by intravenous infusion followed by 40-120 mg LY2090314 by intravenous infusion.
Arm/Group | LY2090314/Pemetrexed/Carboplatin
Number analyzed (Participants) | 41
milligrams (mg) | 40

2. Secondary Outcome: Pharmacokinetic (PK) Parameter: Area Under the Concentration-Time Curve From Time 0 Hour to Infinity (AUC0-∞) of LY2090314
Description: AUC0-∞ was calculated from the area under the concentration versus time curve from time 0 to infinity of LY2090314 when administered alone.
Time Frame: Cycle 1 Day 1 of a 28 day cycle
Population: All participants who received at least 1 dose of LY2090314 and had evaluable AUC0-∞ data, excluding 2 participants (1 in dose groups LY80 and 1 in dose group LY120) who received the wrong dose of LY2090314.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms*hour per milliliter
Groups:
- LY 10/Carb 5 or Carb 6/Pem 500 (Cohorts 1 and 2): * Cycle 1 Day 1 of 28-day cycle: 10 mg LY2090314 by intravenous infusion.
  * Cycle 1 Day 8 of 28-day cycle: 500 mg/m^2 Pem by intravenous infusion followed by AUC 5 (Cohort 1) or AUC 6 (Cohort 2) mg/mL * min Carb by intravenous infusion.
  * Cycle 2 up to Cycle 9: Day 1 of 21-day cycle: 500 mg/m^2 Pem by intravenous infusion followed by AUC 5 (Cohort 1) or AUC 6 (Cohort 2) mg/mL * min Carb by intravenous infusion followed by 10 mg LY2090314 by intravenous infusion.
- LY 40/Carb 6/Pem 500 (Cohorts 4 and 9): * Cycle 1 Day 1 of 28-day cycle: 40 mg LY2090314 by intravenous infusion.
  * Cycle 1 Day 8 of 28-day cycle 500 mg/m^2 Pem by intravenous infusion followed by AUC 6 mg/mL * min Carb by intravenous infusion followed by 40 mg LY2090314 by intravenous infusion.
  * Cycle 2 Day 1 of 21-day cycle: AUC 6 mg/mL * min Carb by intravenous infusion-followed by 500 mg/m^2 Pem by intravenous infusion.
  * Cycle 3 up to Cycle 9: Day 1 of 21-day cycle: 500 mg/m^2 Pem by intravenous infusion followed by AUC 6 mg/mL * min Carb by intravenous infusion followed by 49 mg LY2090314 by intravenous infusion.
  Cohort 9, LY2090314 pretreated with 50 mg ranitidine intravenous.
  Based on I2H-MV-JWYA Protocol Amendment (d) approved 11 March 2010, 50 mg ranitidine was given as a pretreatment to LY2090314 as prophylaxis for stomach pain.
- LY 80/Carb 6/Pem 500 (Cohorts 5 and 7): * Cycle 1 Day 1 of 28-day cycle: 80 mg LY2090314 by intravenous infusion.
  * Cycle 1 Day 8 of 28-day cycle 500 mg/m^2 Pem by intravenous infusion followed by AUC 6 mg/mL * min Carb by intravenous infusion followed by 80 mg LY2090314 by intravenous infusion.
  * Cycle 2 Day 1 of 21-day cycle: AUC 6 mg/mL * min Carb by intravenous infusion followed by 500 mg/m^2 Pem by intravenous infusion.
  * Cycle 3 up to Cycle 10: Day 1 of 21-day cycle: 500 mg/m^2 Pem by intravenous infusion followed by AUC 6 mg/mL * min Carb by intravenous infusion followed by 80 mg LY2090314 by intravenous infusion.
  Cohort 7, LY2090314 pretreated with 50 mg ranitidine intravenous.
  Based on I2H-MV-JWYA Protocol Amendment (d) approved 11 March 2010, 50 mg ranitidine was given as a pretreatment to LY2090314 as prophylaxis for stomach pain.
- LY 120/Carb 6/Pem 500 (Cohort 6): * Cycle 1 Day 1 of 28-day cycle: 120 mg LY2090314 by intravenous infusion.
  * Cycle 1 Day 8 of 28-day cycle 500 mg/m^2 Pem by intravenous infusion followed by AUC 6 mg/mL * min Carb by intravenous infusion followed by 120 mg LY2090314 by intravenous infusion.
  * Cycle 2 Day 1 of 21-day cycle: AUC 6 mg/mL * min Carb by intravenous infusion followed by 500 mg/m^2 by Pem intravenous infusion.
  * Cycle 3 up to Cycle 9: Day 1 of 21-day cycle: 500 mg/m^2 Pem by intravenous infusion followed by AUC 6 mg/mL * min Carb by intravenous infusion followed by 120 mg LY2090314 by intravenous infusion.
- LY 60/Carb 6/Pem 500 + R50 (Cohort 8): * Cycle 1 Day 1 of 28-day cycle: pretreated with 50 mg ranitidine intravenous, 60 mg LY2090314 by intravenous infusion.
  * Cycle 1 Day 8 of 28-day cycle 500 mg/m^2 Pem by intravenous infusion followed by AUC 6mg/mL * min Carb intravenous infusion followed by 50 mg ranitidine intravenous pretreatment and 60 mg LY2090314 by intravenous infusion.
  * Cycle 2 Day 1 of 21-day cycle: AUC 6 mg/mL * min Carb by intravenous infusion followed by 500 mg/m^2 Pem intravenous infusion.
  * Cycle 3 up to Cycle 9: Day 1 of 21-day cycle: 500 mg/m^2 Pem by intravenous infusion followed by AUC 6 mg/mL * min Carb by intravenous infusion followed by pretreatment with 50 mg ranitidine intravenous and 60 mg LY2090314 intravenous infusion.
  Based on I2H-MC-JWYA Protocol Amendment (d) approved 11 March 2010, 50 mg ranitidine was given as a pretreatment to LY2090314 as prophylaxis for stomach pain.
Arm/Group | LY 10/Carb 5 or Carb 6/Pem 500 (Cohorts 1 and 2) | LY 20/Carb 6/Pem 500 (Cohort 3) | LY 40/Carb 6/Pem 500 (Cohorts 4 and 9) | LY 80/Carb 6/Pem 500 (Cohorts 5 and 7) | LY 120/Carb 6/Pem 500 (Cohort 6) | LY 60/Carb 6/Pem 500 + R50 (Cohort 8)
Number analyzed (Participants) | 10 | 5 | 11 | 5 | 3 | 5
nanograms*hour per milliliter | 216 (26.3) | 427 (21.8) | 976 (42.6) | 1870 (76.7) | 3310 (18.7) | 1600 (47.3)

3. Secondary Outcome: PK Parameter: AUC0-∞ of LY2090314 Coadministered With Pemetrexed (Pem) and Carboplatin (Carb)
Description: AUC0-∞ was calculated from the area under the concentration versus time curves of LY2090314 from time zero to infinity when coadministered with Pem and Carb.
Time Frame: Cycle 1 Day 8 of a 28-day cycle or Cycle 2 Day 1 of a 21-day cycle
Population: All participants who received at least 1 dose LY2090314 coadministered with Pem and Carb and had enough samples to allow estimation of AUC0-∞ parameters excluding 2 participants (1 in dose groups LY80 and 1 in dose group LY120) who received the incorrect dose of LY2090314.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms*hour per milliliter
Groups:
- LY 40/Carb 6/Pem 500 (Cohorts 4 and 9): Cycle 1 Day 1 of 28-day cycle: 40 mg LY2090314 by intravenous infusion.
  * Cycle 1 Day 8 of 28-day cycle 500 mg/m^2 Pem by intravenous infusion followed by AUC 6 mg/mL * min Carb by intravenous infusion followed by 40 mg LY2090314 by intravenous infusion.
  * Cycle 2 Day 1 of 21-day cycle: AUC 6 mg/mL * min Carb by intravenous infusion followed by 500 mg/m^2 Pem by intravenous infusion.
  * Cycle 3 up to Cycle 9: Day 1 of 21-day cycle: 500 mg/m^2 Pem by intravenous infusion followed by AUC 6 mg/mL * min Carb by intravenous infusion followed by 40 mg LY2090314 by intravenous infusion.
  Cohort 9, LY2090314 pretreated with 50 mg ranitidine intravenous.
  Based on I2H-MC-JWYa Protocol Amendment (d) approved 11 March 2010, 50 mg ranitidine was given as a pretreatment to LY2090314 as prophylaxis for stomach pain.
- LY 80/Carb 6/Pem 500 (Cohorts 5 and 7): * Cycle 1 Day 1 of 28-day cycle: 80 mg LY2090314 by intravenous infusion.
  * Cycle 1 Day 8 of 28-day cycle 500 mg/m^2 Pem by intravenous infusion followed by AUC 6 mg/mL * min Carb by intravenous infusion followed by 80 mg LY2090314 by intravenous infusion.
  * Cycle 2 Day 1 of 21-day cycle: AUC 6 mg/mL * min Carb by intravenous infusion followed by 500 mg/m^2 Pem by intravenous infusion.
  * Cycle 3 up to Cycle 10: Day 1 of 21-day cycle: 500 mg/m^2 Pem by intravenous infusion followed by AUC 6 mg/mL * min Carb by intravenous infusion followed by 80 mg LY2090314 by intravenous infusion.
  Cohort 7, LY2090314 pretreated with 50 mg ranitidine intravenous.
  Based on I2H-MC-JWYA Protocol Amendment (d) approved 11 March 2010, 50 mg ranitidine was given as a pretreatment to LY2090314 as prophylaxis for stomach pain.
Arm/Group | LY 10/Carb 5 or Carb 6/Pem 500 (Cohorts 1 and 2) | LY 20/Carb 6/Pem 500 (Cohort 3) | LY 40/Carb 6/Pem 500 (Cohorts 4 and 9) | LY 80/Carb 6/Pem 500 (Cohorts 5 and 7) | LY 120/Carb 6/Pem 500 (Cohort 6) | LY 60/Carb 6/Pem 500 + R50 (Cohort 8)
Number analyzed (Participants) | 10 | 4 | 9 | 3 | 1 | 5
nanograms*hour per milliliter | 192 (48.2) | 404 (33.2) | 938 (33.5) | 1830 (7.84) | 2190 (NA) — 1 participant analyzed, therefore, unable to calculate geometric coefficient of variation. | 1570 (36.5)

4. Secondary Outcome: PK Parameter: Maximum Plasma Concentration (Cmax) of LY2090314
Time Frame: Cycle 1 Day 1 of a 28-day cycle
Population: All participants who received at least 1 dose of LY2090314 and had evaluable AUC0-∞ data, excluding 2 participants (1 in dose groups LY80 and 1 in dose group LY120) who received the incorrect dose of LY2090314.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms per milliliter
Groups:
- LY 20/Carb 6/Pem 500 (Cohort 3): * Cycle 1 Day 1 of 28-day cycle: 20 mg LY2090314 by intravenous infusion.
  * Cycle 1 Day 8 of 28-day cycle: 500 mg/m^2 Pem by intravenous infusion followed by AUC 6 mg/mL * min Carb by intravenous infusion.
  * Cycle 2 up to Cycle 9: Day 1 of 21-day cycle: 500 mg/m^2 Pem by intravenous infusion followed by AUC 6 mg/mL * min Carb by intravenous infusion followed by LY2090314 20 mg by intravenous infusion.
- LY 40/Carb 6/Pem 500 (Cohorts 4 and 9 ): Cycle 1 Day 1 of 28-day cycle: 40 mg LY2090314 by intravenous infusion.
  * Cycle 1 Day 8 of 28-day cycle 500 mg/m^2 Pem by intravenous infusion followed by AUC 6 mg/mL * min Carb by intravenous infusion followed by 40 mg LY2090314 by intravenous infusion.
  * Cycle 2 Day 1 of 21-day cycle: AUC 6 mg/mL * min Carb by intravenous infusion followed by 500 mg/m^2 Pem by intravenous infusion.
  * Cycle 3 up to Cycle 9: Day 1 of 21-day cycle: 500 mg/m^2 Pem by intravenous infusion followed by AUC 6 mg/mL * min Carb by intravenous infusion followed by 49 mg LY2090314 by intravenous infusion.
  Cohort 9, LY2090314 pretreated with 50 mg ranitidine IV. Based on I2H-MC-JWYA Protocol Amendment (d) approved 11 March 2010, 50 mg ranitidine was given as a pretreatment to LY2090314 as prophylaxis for stomach pain.
- LY 80/Carb 6/Pem 500 (Cohorts 5 and 7: * Cycle 1 Day 1 of 28-day cycle: 80 mg LY2090314 by intravenous infusion.
  * Cycle 1 Day 8 of 28-day cycle 500 mg/m^2 Pem by intravenous infusion followed by AUC 6 mg/mL * min Carb by intravenous infusion followed by 80 mg LY2090314 by intravenous infusion.
  * Cycle 2 Day 1 of 21-day cycle: AUC 6 mg/mL * min Carb by intravenous infusion followed by 500 mg/m^2 Pem by intravenous infusion.
  * Cycle 3 up to Cycle 10: Day 1 of 21-day cycle: 500 mg/m^2 Pem by intravenous infusion followed by AUC 6 mg/mL * min Carb by intravenous infusion followed by 80 mg LY2090314 by intravenous infusion.
  Cohort 7, LY2090314 pretreated with 50 mg ranitidine IV.
  Based on I2H-MC-JWYA Protocol Amendment (d) approved 11 March 2010, 50 mg ranitidine was given as a pretreatment to LY2090314 as prophylaxis for stomach pain.
- LY 60/Carb 6/Pem 500 + R50 (Cohort 8): * Cycle 1 Day 1 of 28-day cycle: pretreated with 50 mg ranitidine intravenous, 60 mg LY2090314 by IV infusion.
  * Cycle 1 Day 8 of 28-day cycle 500 mg/m^2 Pem by intravenous infusion followed by AUC 6mg/mL * min Carb intravenous infusion followed by 50 mg ranitidine intravenous pretreatment and 60 mg LY2090314 by intravenous infusion.
  * Cycle 2 Day 1 of 21-day cycle: AUC 6 mg/mL * min Carb by intravenous infusion followed by 500 mg/m^2 Pem intravenous infusion.
  * Cycle 3 up to Cycle 9: Day 1 of 21-day cycle: 500 mg/m^2 Pem by intravenous infusion followed by AUC 6 mg/mL * min Carb by intravenous infusion followed by pretreatment with 50 mg ranitidine intravenous and 60 mg LY2090314 intravenous infusion.
  Based on I2H-MC-JWYA Protocol Amendment (d) approved 11 March 2010, 50 mg ranitidine was given as a pretreatment to LY2090314 as prophylaxis for stomach pain.
Arm/Group | LY 10/Carb 5 or Carb 6/Pem 500 (Cohorts 1 and 2) | LY 20/Carb 6/Pem 500 (Cohort 3) | LY 40/Carb 6/Pem 500 (Cohorts 4 and 9 ) | LY 80/Carb 6/Pem 500 (Cohorts 5 and 7 | LY 120/Carb 6/Pem 500 (Cohort 6) | LY 60/Carb 6/Pem 500 + R50 (Cohort 8)
Number analyzed (Participants) | 10 | 5 | 11 | 5 | 3 | 5
nanograms per milliliter | 122 (21.5) | 246 (29.0) | 603 (47.7) | 898 (50.5) | 1700 (63.2) | 881 (53.3)

5. Secondary Outcome: PK Parameter: Maximum Plasma Concentration (Cmax) of LY2090314 Coadministered With Pemetrexed (Pem) and Carboplatin (Carb)
Time Frame: Cycle 1 Day 8 of a 28-day cycle or Cycle 2 Day 1 of a 21-day cycle
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms per milliliter
Groups:
- LY 40/Carb 6/Pem 500 (Cohorts 4 and 9): Cycle 1 Day 1 of 28-day cycle: 40 mg LY2090314 by intravenous infusion.
  * Cycle 1 Day 8 of 28-day cycle 500 mg/m^2 Pem by intravenous infusion followed by AUC 6 mg/mL * min Carb by intravenous infusion followed by 40 mg LY2090314 by intravenous infusion.
  * Cycle 2 Day 1 of 21-day cycle: AUC 6 mg/mL * min Carb by intravenous infusion followed by 500 mg/m^2 Pem by intravenous infusion.
  * Cycle 3 up to Cycle 10: Day 1 of 21-day cycle: 500 mg/m^2 Pem by intravenous infusion followed by AUC 6 mg/mL * min Carb by intravenous infusion followed by 40 mg LY2090314 by intravenous infusion.
  Cohort 9, LY2090314 pretreated with 50 mg ranitidine intravenous.
  Based on I2H-MC-JWYA Protocol Amendment (d) approved 11 March 2010, 50 mg ranitidine was given as a pretreatment to LY2090314 as prophylaxis for stomach pain.
- LY 80/Carb 6/Pem 500 (Cohorts 5 and 7): * Cycle 1 Day 1 of 28-day cycle: 80 mg LY2090314 by intravenous infusion.
  * Cycle 1 Day 8 of 28-day cycle 500 mg/m^2 Pem by intravenous infusion followed by AUC 6 mg/mL * min Carb by intravenous infusion followed by 80 mg LY2090314 by intravenous infusion.
  * Cycle 2 Day 1 of 21-day cycle: AUC 6 mg/mL * min Carb by intravenous infusion followed by 500 mg/m^2 Pem by intravenous infusion.
  * Cycle 3 up to Cycle 10: Day 1 of 21-day cycle: 500 mg/m^2 Pem by intravenous infusion followed by AUC 6 mg/mL * min Carb by intravenous infusion followed by 80 mg LY2090314 by intravenous infusion.
  Cohort 7, LY2090314 pretreated with 50 mg ranitidine IV.
  Based on I2H-MC-JWYA Protocol Amendment (d) approved 11 March 2010, 50 mg ranitidine was given as a pretreatment to LY2090314 as prophylaxis for stomach pain.
- LY 60/Carb 6/Pem 500 + R50 (Cohort 8): * Cycle 1 Day 1 of 28-day cycle: pretreated with 50 mg ranitidine intravenous, 60 mg LY2090314 by intravenous infusion.
  * Cycle 1 Day 8 of 28-day cycle 500 mg/m^2 Pem by intravenous infusion followed by AUC 6mg/mL * min Carb intravenous infusion followed by 50 mg ranitidine intravenous pretreatment and 60 mg LY2090314 by intravenous infusion.
  * Cycle 2 Day 1 of 21-day cycle: AUC 6 mg/mL * min Carb by intravenous infusion followed by 500 mg/m^2 Pem intravenous infusion.
  * Cycle 3 up to Cycle 9: Day 1 of 21-day cycle: 500 mg/m^2 Pem by intravenous infusion followed by AUC 6 mg/mL * min Carb by intravenous infusion followed by pretreatment with 50 mg ranitidine intravenous and 60 mg LY2090314 intravenous infusion.
  Based on I2H-MC_JWYA Protocol Amendment (d) approved 11 March 2010, 50 mg ranitidine was given as a pretreatment to LY2090314 as prophylaxis for stomach pain.
Arm/Group | LY 10/Carb 5 or Carb 6/Pem 500 (Cohorts 1 and 2) | LY 20/Carb 6/Pem 500 (Cohort 3) | LY 40/Carb 6/Pem 500 (Cohorts 4 and 9) | LY 80/Carb 6/Pem 500 (Cohorts 5 and 7) | LY 120/Carb 6/Pem 500 (Cohort 6) | LY 60/Carb 6/Pem 500 + R50 (Cohort 8)
Number analyzed (Participants) | 10 | 4 | 9 | 3 | 1 | 5
nanograms per milliliter | 106 (57.5) | 271 (62.5) | 657 (44.1) | 1150 (27.8) | 768 (NA) — 1 participant analyzed, therefore, unable to calculate geometric coefficient of variation. | 1040 (48.2)

6. Secondary Outcome: Number of Participants With Best Overall Tumor Response
Description: Best overall observed tumor response at any point during the study until disease progression/recurrence defined using Response Evaluation Criteria In Solid Tumors (RECIST) criteria. Complete Response (CR) was defined as the disappearance of all target and non-target lesions and any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 millimeter (mm) and normalization of tumor marker level of non-target lesions; Partial Response (PR) was defined as at least 30% decrease in sum of longest diameter of target lesions; Progressive Disease (PD) was defined as at least 20% increase in sum of longest diameter of target lesions and minimum 5 mm increase over nadir; Stable Disease (SD) was defined as small changes that did not meet above criteria.
Time Frame: Baseline up to Cycle 9 (Cycle 1 was 28 days, Cycles 2 to 9 were 21 days)
Population: Analysis population: all participants who received at least 1 dose of study drug and had tumor response assessment.
Measure: Number; unit: participants
Groups:
- LY 80/Carb 6/Pem 500 + R50 (Cohort 7): * Cycle 1 Day 1 of 28-day cycle: pretreated with 50 mg ranitidine intravenous, 80 mg LY2090314 by intravenous infusion.
  * Cycle 1 Day 8 of 28-day cycle 500 mg/m^2 Pem by intravenous infusion followed by AUC 6mg/mL * min Carb intravenous infusion followed by 50 mg ranitidine intravenous pretreatment and 80 mg LY2090314 by intravenous infusion.
  * Cycle 2 Day 1 of 21-day cycle: AUC 6 mg/mL * min Carb by intravenous infusion followed by 500 mg/m^2 Pem intravenous infusion.
  * Cycle 3 up to Cycle 10: Day 1 of 21-day cycle: 500 mg/m^2 Pem by intravenous infusion followed by AUC 6 mg/mL * min Carb by intravenous infusion followed by 50 mg ranitidine intravenous pretreatment and 80 mg LY2090314 IV infusion.
  Based on I2H-MC-JWYA Protocol Amendment (d) approved 11 March 2010, 50 mg ranitidine was given as a pretreatment to LY2090314 as prophylaxis for stomach pain.
- LY 40/Carb 6/Pem 500 + R50 (Cohort 9): * Cycle 1 Day 1 of 28-day cycle: pretreated with 50 mg ranitidine intravenous, 40 mg LY2090314 by intravenous infusion.
  * Cycle 1 Day 8 of 28-day cycle 500 mg/m^2 Pem by intravenous infusion followed by AUC 6mg/mL * min Carb intravenous infusion followed by 50 mg ranitidine intravenous pretreatment and 40 mg LY2090314 by intravenous infusion.
  * Cycle 2 Day 1 of 21-day cycle: AUC 6 mg/mL * min Carb by intravenous infusion followed by 500 mg/m^2 intravenous Pem infusion.
  * Cycle 3 up to Cycle 9: Day 1 of 21-day cycle: 500 mg/m^2 Pem by intravenous infusion followed by AUC 6 mg/mL * min by Carb intravenous infusion followed by 50 mg ranitidine intravenous pretreatment and 40 mg LY2090314 intravenous infusion.
  Based on I2H-MC-JWYA Protocol Amendment (d) approved 11 March 2010, 50 mg ranitidine was given as a pretreatment to LY2090314 as prophylaxis for stomach pain.
Arm/Group | LY 10/Carb 5/Pem 500 (Cohort 1) | LY 10/Carb 6/Pem 500 (Cohort 2) | LY 20/Carb 6/Pem 500 (Cohort 3) | LY 40/Carb 6/Pem 500 (Cohort 4) | LY 80/Carb 6/Pem 500 (Cohort 5) | LY 120/Carb 6/Pem 500 (Cohort 6) | LY 80/Carb 6/Pem 500 + R50 (Cohort 7) | LY 60/Carb 6/Pem 500 + R50 (Cohort 8) | LY 40/Carb 6/Pem 500 + R50 (Cohort 9)
Number analyzed (Participants) | 3 | 7 | 5 | 7 | 3 | 4 | 2 | 5 | 5
participants
  CR | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  PR | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 1 | 0
  SD | 2 | 4 | 2 | 2 | 0 | 0 | 1 | 1 | 2
  PD | 0 | 2 | 1 | 3 | 1 | 0 | 0 | 2 | 2
  Unknown (discontinued before response assessment) | 1 | 1 | 1 | 0 | 2 | 0 | 0 | 0 | 1

7. Secondary Outcome: Pharmacokinetic (PK) Parameter: Area Under the Concentration-Time Curve From Time 0 Hour to Infinity (AUC0-∞) of Pemetrexed (Pem)
Description: AUC0-∞ was calculated from the area under the concentration versus time curves of Pem given as a single dose with Carb (doublet therapy) and when co-administered with Carb and LY2090314 (triplet therapy).
Time Frame: Cycle 1 Day 8 of 28-day cycle and Cycle 2 up to Cycle 10 Day 1 of 21-day cycle
Population: All participants who were treated with Pem and Carb (doublet therapy) or who were treated with Pem, Carb and LY2090314 (triplet therapy) and had evaluable AUC0-∞ Pem data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours*nanograms/milliliter/ milligram
Groups:
- Pemetrexed (Doublet Therapy): Pem with Carb
  * Participants in Cohorts 1, 2 and 3 were administered 500 mg/m^2 Pem and AUC 5 or AUC 6 mg/mL * min Carb on Cycle 1, Day 8 of 28-day cycle by intravenous infusion.
  * Participants in Cohorts 4 through 9 were administered 500 mg/m^2 Pem and AUC 6 mg/mL * min Carb by intravenous infusion on Cycle 2 Day 1 of 21-day cycle
- Pemetrexed (Triplet Therapy): Pem with Carb and LY2090314
  * Participants in Cohorts 1, 2 and 3 were administered 500 mg/m^2 Pem by intravenous infusion followed by AUC 5 or AUC 6 mg/mL * min Carb by intravenous infusion followed by 10 mg up to 20 mg LY2090314 by intravenous infusion on Cycle 2 up to Cycle 10: Day 1 of 21-day cycle.
  * Participants in Cohorts 4 through 9 were administered 500 mg/m^2 Pem and AUC 6 mg/mL * min Carb by intravenous infusion followed by 40 mg up to 120 mg of LY2090314 by intravenous infusion on Cycle 1, Day 8 of 28-day cycle and Cycle 3 up to Cycle 10: Day 1 of 21-day cycle.
  Based on I2H-MC-JWYA Protocol Amendment (D) approved 11 March 2010, 50 mg ranitidine was given as a pretreatment to LY2090314 as prophylaxis for stomach pain to participants in Cohorts 7, 8 and 9.
Arm/Group | Pemetrexed (Doublet Therapy) | Pemetrexed (Triplet Therapy)
Number analyzed (Participants) | 33 | 36
hours*nanograms/milliliter/ milligram | 212 (34.4) | 202 (37.5)

8. Secondary Outcome: PK Parameter: Maximum Plasma Concentration (Cmax) of Pemetrexed (Pem)
Description: Cmax of Pem given as a single dose with Carb (doublet therapy) and when coadministered with Carb and LY2090314 (triplet therapy).
Time Frame: Cycle 1 Day 8 of 28-day cycle and Cycle 2 up to Cycle 10 Day 1 of 21-day cycle
Population: All participants who were treated with Pem and Carb (doublet therapy) or who were treated with Pem, Carb and LY2090314 (triplet therapy) and had evaluable Cmax Pem data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter per milligram
Groups:
- Pemetrexed (Triplet Therapy): Pem with Carb and LY2090317
  * Participants in Cohorts 1, 2 and 3 were administered 500 mg/m^2 Pem by intravenous infusion followed by AUC 5 or AUC 6 mg/mL * min Carb by intravenous infusion followed by 10 mg up to 20 mg LY2090314 by intravenous infusion on Cycle 2 up to Cycle 10: Day 1 of 21-day cycle.
  * Participants in Cohorts 4 through 9 were administered 500 mg/m^2 Pem and AUC 6 mg/mL * min Carb by intravenous infusion followed by 40 mg up to 120 mg of LY2090314 by intravenous infusion on Cycle 1, Day 8 of 28-day cycle and Cycle 3 up to Cycle 10: Day 1 of 21-day cycle.
  Based on I2H-MC-JWYA Protocol Amendment (d) approved 11 March 2010, 50 mg ranitidine was given as a pretreatment to LY2090314 as prophylaxis for stomach pain to participants in Cohorts 7, 8 and 9.
Arm/Group | Pemetrexed (Doublet Therapy) | Pemetrexed (Triplet Therapy)
Number analyzed (Participants) | 33 | 36
nanogram per milliliter per milligram | 109 (38.0) | 108 (43.1)

9. Secondary Outcome: PK Parameter: AUC0-∞ of Free Carboplatin (Carb)
Description: AUC0-∞ of free Carb was calculated from the area under the concentration versus time curves of Carb given as a single dose with Pem (doublet therapy) and when co-administered with Pem and LY2090314 (triplet therapy).
Time Frame: Cycle 1 Day 8 of 28-day cycle and Cycle 2 up to Cycle 9: Day 1 of 21-day cycle
Population: All participants who were treated with Pem and Carb (doublet therapy) or Pem, Carb and LY2090314 (triplet therapy) and who had evaluable Carb AUC0-∞ data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours*nanograms per milliliter per mg
Groups:
- Carboplatin (Doublet Therapy): Carb and Pem
  * Participants in Cohorts 1, 2 and 3 were administered 500 mg/m^2 Pem and AUC 5 or AUC 6 mg/mL * min Carb on Cycle 1, Day 8 of 28-day cycle by intravenous infusion.
  * Participants in Cohorts 4 through 9 were administered 500 mg/m^2 Pem and AUC 6 mg/mL * min Carb by intravenous infusion on Cycle 2 Day 1 of 21-day cycle
- Carboplatin (Triplet Therapy): Carb with Pem and LY2090314
  * Participants in Cohorts 1, 2 and 3 were administered 500 mg/m^2 Pem by intravenous infusion followed by AUC 5 or AUC 6 mg/mL * min Carb by intravenous infusion followed by 10 mg up to 20 mg LY2090314 by intravenous infusion on Cycle 2 up to Cycle 9: Day 1 of 21-day cycle.
  * Participants in Cohorts 4 through 9 were administered 500 mg/m^2 Pem and AUC 6 mg/mL * min Carb by intravenous infusion followed by 40 mg up to 120 mg of LY2090314 by intravenous infusion on Cycle 1, Day 8 of 28-day cycle and Cycle 3 up to Cycle 9: Day 1 of 21-day cycle.
  Based on I2H-MC-JWYA Protocol Amendment (d) approved 11 March 2010, 50 mg ranitidine was given as a pretreatment to LY2090314 as prophylaxis for stomach pain to participants in Cohorts 7, 8 and 9.
Arm/Group | Carboplatin (Doublet Therapy) | Carboplatin (Triplet Therapy)
Number analyzed (Participants) | 32 | 35
hours*nanograms per milliliter per mg | 81.6 (41.8) | 88.1 (49.2)

10. Secondary Outcome: PK Parameter: Cmax of Free Carboplatin
Description: Cmax of free Carb given as a single dose with Pem (doublet therapy) and when co-administered with Pem and LY2090314 (triplet therapy).
Time Frame: Cycle 1, Day 8 of 28-day cycle and Cycle 2 up to Cycle 9: Day 1 of 21-day cycle
Population: All participants who were treated with Pem and Carb (doublet therapy) or who were treated with Pem, Carb and LY2090314 (triplet therapy) and had evaluable Carb Cmax data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms/milliliter/milligram
Groups:
- Carboplatin (Triplet Therapy): Carb and Pem with LY2090314
  * Participants in Cohorts 1, 2 and 3 were administered 500 mg/m^2 Pem by intravenous infusion followed by AUC 5 or AUC 6 mg/mL * min Carb by intravenous infusion followed by 10 mg up to 20 mg LY2090314 by intravenous infusion on Cycle 2 up to Cycle 9: Day 1 of 21-day cycle.
  * Participants in Cohorts 4 through 9 were administered 500 mg/m^2 Pem and AUC 6 mg/mL * min Carb by intravenous infusion followed by 40 mg up to 120 mg of LY2090314 by intravenous infusion on Cycle 1, Day 8 of 28-day cycle and Cycle 3 up to Cycle 10: Day 1 of 21-day cycle.
  Based on I2H-MC-JWYA Protocol Amendment (d) approved 11 March 2010, 50 mg ranitidine was given as a pretreatment to LY2090314 as prophylaxis for stomach pain to participants in Cohorts 7, 8 and 9.
Arm/Group | Carboplatin (Doublet Therapy) | Carboplatin (Triplet Therapy)
Number analyzed (Participants) | 32 | 35
nanograms/milliliter/milligram | 24.0 (43.9) | 25.5 (46.0)

11. Secondary Outcome: Pharmacodynamic (PD) Changes in Beta-Catenin (β-catenin)
Description: PD change from baseline to endpoint (up to Cycle 9) in β-catenin levels in peripheral blood mononuclear cells (PBMCs) following the administration of LY2090314 given alone and in combination with Pem and Carb. This outcome measure was not analyzed due to insufficient data.
Time Frame: Baseline, Cycle 1 , Day 1 of a 28-day cycle and Cycle 2 up to Cycle 9: Day 1 of 21-day cycles
Population: There was insufficient data from participants who received at least 1 dose of LY2090314 to perform β-catenin modeling, thus zero participants were analyzed.
Groups:
- LY 10/Carb 5/Pem 500 (Cohort 1): * Cycle 1 Day 1 of 28-day cycle: 10 mg LY2090314 by intravenous infusion.
  * Cycle 1 Day 8 of 28-day cycle: 500 mg/m^2 Pem by intravenous infusion followed by AUC 5 mg/mL * min Carb by IV infusion.
  * Cycle 2 up to Cycle 9: Day 1 of 21-day cycle: 500 mg/m^2 Pem by intravenous infusion followed by AUC 5 mg/mL * min Carb by intravenous infusion followed by 10 mg LY2090314 by intravenous infusion.
- LY 10/Carb 6/Pem 500 (Cohort 2): * Cycle 1 Day 1 of 28-day cycle: 10 mg LY2090314 by IV infusion.
  * Cycle 1 Day 8 of 28-day cycle: 500 mg/m^2 Pem by intravenous infusion followed by AUC 6 mg/mL * min Carb by intravenous infusion.
  * Cycle 2 up to Cycle 9: Day 1 of 21-day cycle: 500 mg/m^2 Pem by intravenous infusion followed by AUC 6 mg/mL * min Carb by intravenous infusion followed by 10 mg LY2090314 by intravenous infusion.
- LY 20/Carb 6/Pem 500 (Cohort 3): * Cycle 1 Day 1 of 28-day cycle: 20 mg LY2090314 by intravenous infusion.
  * Cycle 1 Day 8 of 28 -ay cycle: 500 mg/m^2 Pem by intravenous infusion followed by AUC 6 mg/mL * min Carb by intravenous infusion.
  * Cycle 2 up to Cycle 9: Day 1 of 21-day cycle: 500 mg/m^2 Pem by intravenous infusion followed by AUC 6 mg/mL * min Carb by intravenous infusion followed by 20 mg LY2090314 by intravenous infusion.
- LY 120/Carb 6/Pem 500 (Cohort 6): * Cycle 1 Day 1 of 28-day cycle: 120 mg LY2090314 mg by intravenous infusion.
  * Cycle 1 Day 8 of 28-day cycle 500 mg/m^2 Pem by intravenous infusion followed by AUC 6 mg/mL * min Carb by intravenous infusion followed by 120 mg LY2090314 by intravenous infusion.
  * Cycle 2 Day 1 of 21-day cycle: AUC 6 mg/mL * min Carb by intravenous infusion followed by 500 mg/m^2 Pem by intravenous infusion.
  * Cycle 3 up to Cycle 9: Day 1 of 21-day cycle: 500 mg/m^2 Pem by intravenous infusion followed by AUC 6 mg/mL * min Carb by intravenous infusion followed by 120 mg LY2090314 by intravenous infusion.
- LY 80/Carb 6/Pem 500 + R50 (Cohort 7): * Cycle 1 Day 1 of 28-day cycle: pretreated with 50 mg ranitidine intravenous, 80 mg LY2090314 by intravenous infusion.
  * Cycle 1 Day 8 of 28-day cycle 500 mg/m^2 Pem by intravenous infusion followed by AUC 6 mg/mL * min Carb intravenous infusion followed by 50 mg ranitidine intravenous pretreatment and 80 mg LY2090314 by intravenous infusion.
  * Cycle 2 Day 1 of 21-day cycle: AUC 6 mg/mL * min Carb by intravenous infusion followed by 500 mg/m^2 Pem intravenous infusion.
  * Cycle 3 up to Cycle 10: Day 1 of 21-day cycle: 500 mg/m^2 Pem by intravenous infusion followed by AUC 6 mg/mL * min Carb by intravenous infusion followed by 50 mg ranitidine intravenous pretreatment and 80 mg LY2090314 intravenous infusion.
  Based on I2H-MC-JWYA Protocol Amendment (d) approved 11 March 2010, 50 mg ranitidine was given as a pretreatment to LY2090314 as prophylaxis for stomach pain.
- LY 60/Carb 6/Pem 500 + R50 (Cohort 8): * Cycle 1 Day 1 of 28-day cycle: pretreated with 50 mg ranitidine intravenous, 60 mg LY2090314 by intravenous infusion.
  * Cycle 1 Day 8 of 28-day cycle 500 mg/m^2 Pem by intravenous infusion followed by AUC 6mg/mL * min Carb intravenous infusion followed by 50 mg ranitidine intravenous pretreatment and 60 mg LY2090314 by intravenous infusion.
  * Cycle 2 Day 1 of 21-day cycle: AUC 6 mg/mL * min Carb by intravenous infusion followed by 500 mg/m^2 Pem intravenous infusion.
  * Cycle 3 up to Cycle 9: Day 1 of 21-day cycle: 500 mg/m^2 Pem by intravenous infusion followed by AUC 6 mg/mL * min Carb by intravenous infusion followed by 50 mg ranitidine IV pretreatment and 60 mg LY2090314 intravenous infusion.
  Based on I2H-MC-JWYA Protocol Amendment (d) approved 11 March 2010, 50 mg ranitidine was given as a pretreatment to LY2090314 as prophylaxis for stomach pain.
Arm/Group | LY 10/Carb 5/Pem 500 (Cohort 1) | LY 10/Carb 6/Pem 500 (Cohort 2) | LY 20/Carb 6/Pem 500 (Cohort 3) | LY 40/Carb 6/Pem 500 (Cohort 4) | LY 80/Carb 6/Pem 500 (Cohort 5) | LY 120/Carb 6/Pem 500 (Cohort 6) | LY 80/Carb 6/Pem 500 + R50 (Cohort 7) | LY 60/Carb 6/Pem 500 + R50 (Cohort 8) | LY 40/Carb 6/Pem 500 + R50 (Cohort 9)
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Groups:
- LY 10/Carb 5/Pem 500 (Cohort 1): * Cycle 1 Day 1 of 28 day cycle: 10 mg LY2090314 administered by intravenous infusion.
  * Cycle 1 Day 8 of 28 day cycle: 500 mg/m^2 Pem administered by intravenous infusion followed by AUC 5 mg/mL * min Carb administered by intravenous infusion.
  * Cycle 2 up to Cycle 9: Day 1 of 21 day cycle: 500 mg/m^2 Pem administered by intravenous infusion followed by AUC 5 mg/mL * min Carb administered by intravenous infusion followed by 10 mg LY2090314 administered by intravenous infusion.
- LY 10/Carb 6/Pem 500 (Cohort 2): * Cycle 1 Day 1 of 28 day cycle: 10 mg LY2090314 by intravenous infusion.
  * Cycle 1 Day 8 of 28 day cycle: 500 mg/m^2 by Pem intravenous infusion followed by AUC 6 mg/mL * min Carb by intravenous infusion.
  * Cycle 2 up to Cycle 9: Day 1 of 21 day cycle: 500 mg/m^2 Pem by intravenous infusion followed by AUC 6 mg/mL * min Carb by intravenous infusion followed by 10 mg LY2090314 by intravenous infusion.
- LY 20/Carb 6/Pem 500 (Cohort 3): * Cycle 1 Day 1 of 28 day cycle: 20 mg LY2090314 by intravenous infusion.
  * Cycle 1 Day 8 of 28 day cycle: 500 mg/m^2 Pem by intravenous infusion followed by AUC 6 mg/mL * min Carb by intravenous infusion.
  * Cycle 2 up to Cycle 9: Day 1 of 21 day cycle: 500 mg/m^2 Pem by intravenous infusion followed by AUC 6 mg/mL * min Carb by intravenous infusion followed by 20 mg LY2090314 by intravenous infusion.
- LY 40/Carb 6/Pem 500 (Cohort 4): * Cycle 1 Day 1 of 28 day cycle: 40 mg LY2090314 by intravenous infusion.
  * Cycle 1 Day 8 of 28 day cycle: 500 mg/m^2 Pem by intravenous infusion followed by AUC 6 mg/mL * min Carb by intravenous infusion followed by 40 mg LY2090314 by intravenous infusion.
  * Cycle 2 Day 1 of 21 day cycle: AUC 6 mg/mL * min Carb by intravenous infusion followed by 500 mg/m^2 Pem by intravenous infusion.
  * Cycle 3 up to Cycle 9: Day 1 of 21 day cycle: 500 mg/m^2 Pem by intravenous infusion followed by AUC 6 mg/mL * min Carb by intravenous infusion followed by 40 mg LY2090314 by intravenous infusion.
- LY 80/Carb 6/Pem 500 (Cohort 5): * Cycle 1 Day 1 of 28 day cycle: 80 mg LY2090314 by intravenous infusion.
  * Cycle 1 Day 8 of 28 day cycle: 500 mg/m^2 Pem by intravenous infusion followed by AUC 6 mg/mL * min Carb by intravenous infusion followed by 80 mg LY2090314 by intravenous infusion.
  * Cycle 2 Day 1 of 21 day cycle: AUC 6 mg/mL * min Carb by intravenous infusion followed by 500 mg/m^2 Pem by intravenous infusion.
  * Cycle 3 up to Cycle 9: Day 1 of 21 day cycle: 500 mg/m^2 Pem by intravenous infusion followed by AUC 6 mg/mL * min Carb by intravenous infusion followed by 80 mg LY2090314 by intravenous infusion.
- LY 120/Carb 6/Pem 500 (Cohort 6): * Cycle 1 Day 1 of 28 day cycle: 120 mg LY2090314 by intravenous infusion.
  * Cycle 1 Day 8 of 28 day cycle: 500 mg/m^Pem by intravenous infusion followed by AUC 6 mg/mL * min Carb by intravenous infusion followed by 120 mg LY2090314 by intravenous infusion.
  * Cycle 2 Day 1 of 21 day cycle: AUC 6 mg/mL * min Carb by intravenous infusion followed by 500 mg/m^2 Pem by intravenous infusion.
  * Cycle 3 up to Cycle 9: Day 1 of 21 day cycle: 500 mg/m^2 Pem by intravenous infusion followed by AUC 6 mg/mL * min Carb by intravenous infusion followed by 120 mg LY2090314 by intravenous infusion.
- LY 80/Carb 6/Pem 500 + R50 (Cohort 7): * Cycle 1 Day 1 of 28 day cycle: pretreated with 50 mg ranitidine intravenous, 80 mg LY2090314 by intravenous infusion.
  * Cycle 1 Day 8 of 28 day cycle: 500 mg/m^2 Pem by intravenous infusion followed by AUC 6mg/mL * min Carb intravenous infusion followed by 50 mg ranitidine intravenous pretreatment and 80 mg LY2090314 by intravenous infusion.
  * Cycle 2 Day 1 of 21 day cycle: AUC 6 mg/mL * min Carb by intravenous infusion followed by 500 mg/m^2 Pem intravenous infusion.
  * Cycle 3 up to Cycle 9: Day 1 of 21 day cycle: 500 mg/m^2 Pem by intravenous infusion followed by AUC 6 mg/mL * min Carb by intravenous infusion followed by 50 mg ranitidine intravenous pretreatment and 80 mg LY2090314 intravenous infusion.
  Based on I2H-MV-JWYA Protocol Amendment (d) approved 11 March 2010, 50 mg ranitidine was given as a pretreatment to LY2090314 as prophylaxis for stomach pain.
- LY 60/Carb 6/Pem 500 + R50 (Cohort 8): * Cycle 1 Day 1 of 28 day cycle: pretreated with 50 mg ranitidine intravenous, 60 mg LY2090314 by intravenous infusion.
  * Cycle 1 Day 8 of 28 day cycle: 500 mg/m^2 Pem by intravenous infusion followed by AUC 6mg/mL * min Carb intravenous infusion followed by 50 mg ranitidine intravenous pretreatment and 60 mg LY2090314 by intravenous infusion.
  * Cycle 2 Day 1 of 21 day cycle: AUC 6 mg/mL * min Carb by intravenous infusion followed by 500 mg/m^2 Pem intravenous infusion.
  * Cycle 3 up to Cycle 9: Day 1 of 21 day cycle: 500 mg/m^2 Pem by intravenous infusion followed by AUC 6 mg/mL * min Carb by intravenous infusion followed by 50 mg ranitidine intravenous pretreatment and 60 mg LY2090314 intravenous infusion.
  Based on I2H-MV-JWYA Protocol Amendment (d) approved 11 March 2010, 50 mg ranitidine was given as a pretreatment to LY2090314 as prophylaxis for stomach pain.
- LY 40/Carb 6/Pem 500 + R50 (Cohort 9): * Cycle 1 Day 1 of 28 day cycle: pretreated with 50 mg ranitidine intravenous, 40 mg LY2090314 by intravenous infusion.
  * Cycle 1 Day 8 of 28 day cycle: 500 mg/m^2 Pem by intravenous infusion followed by AUC 6mg/mL * min Carb intravenous infusion followed by 50 mg ranitidine intravenous pretreatment and 40mmg LY2090314 40 mg by intravenous infusion.
  * Cycle 2 Day 1 of 21 day cycle: AUC 6 mg/mL * min Carb by intravenous infusion followed by 500 mg/m^2 Pem intravenous infusion.
  * Cycle 3 up to Cycle 9: Day 1 of 21 day cycle: 500 mg/m^2 Pem by intravenous infusion followed by AUC 6 mg/mL * min Carb by intravenous infusion followed by 50 mg ranitidine intravenous pretreatment and 40 mg LY2090314 intravenous infusion.
  Based on I2H-MV-JWYA Protocol Amendment (d) approved 11 March 2010, 50 mg ranitidine was given as a pretreatment to LY2090314 as prophylaxis for stomach pain.
Arm/Group | LY 10/Carb 5/Pem 500 (Cohort 1) | LY 10/Carb 6/Pem 500 (Cohort 2) | LY 20/Carb 6/Pem 500 (Cohort 3) | LY 40/Carb 6/Pem 500 (Cohort 4) | LY 80/Carb 6/Pem 500 (Cohort 5) | LY 120/Carb 6/Pem 500 (Cohort 6) | LY 80/Carb 6/Pem 500 + R50 (Cohort 7) | LY 60/Carb 6/Pem 500 + R50 (Cohort 8) | LY 40/Carb 6/Pem 500 + R50 (Cohort 9)
Serious Adverse Events (participants affected / at risk) | 1/3 | 3/7 | 3/5 | 2/7 | 1/3 | 1/4 | 1/2 | 0/5 | 1/5
Other Adverse Events (participants affected / at risk) | 3/3 | 7/7 | 5/5 | 7/7 | 3/3 | 3/4 | 2/2 | 5/5 | 5/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LY 10/Carb 5/Pem 500 (Cohort 1) (N=3) | LY 10/Carb 6/Pem 500 (Cohort 2) (N=7) | LY 20/Carb 6/Pem 500 (Cohort 3) (N=5) | LY 40/Carb 6/Pem 500 (Cohort 4) (N=7) | LY 80/Carb 6/Pem 500 (Cohort 5) (N=3) | LY 120/Carb 6/Pem 500 (Cohort 6) (N=4) | LY 80/Carb 6/Pem 500 + R50 (Cohort 7) (N=2) | LY 60/Carb 6/Pem 500 + R50 (Cohort 8) (N=5) | LY 40/Carb 6/Pem 500 + R50 (Cohort 9) (N=5)
Angina pectoris (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pseudomembranous colitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Panic attack (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LY 10/Carb 5/Pem 500 (Cohort 1) (N=3) | LY 10/Carb 6/Pem 500 (Cohort 2) (N=7) | LY 20/Carb 6/Pem 500 (Cohort 3) (N=5) | LY 40/Carb 6/Pem 500 (Cohort 4) (N=7) | LY 80/Carb 6/Pem 500 (Cohort 5) (N=3) | LY 120/Carb 6/Pem 500 (Cohort 6) (N=4) | LY 80/Carb 6/Pem 500 + R50 (Cohort 7) (N=2) | LY 60/Carb 6/Pem 500 + R50 (Cohort 8) (N=5) | LY 40/Carb 6/Pem 500 + R50 (Cohort 9) (N=5)
Anaemia (Blood and lymphatic system disorders) | 2 (3) | 6 (8) | 5 (5) | 5 (5) | 2 (3) | 0 (0) | 1 (1) | 4 (4) | 3 (5)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 4 (4) | 1 (1) | 3 (8) | 2 (3) | 0 (0) | 1 (2) | 2 (2) | 1 (2)
Lymphopenia (Blood and lymphatic system disorders) | 0 (0) | 4 (4) | 1 (1) | 3 (4) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 4 (7) | 2 (6) | 5 (14) | 3 (4) | 0 (0) | 1 (1) | 3 (6) | 2 (4)
Thrombocytopenia (Blood and lymphatic system disorders) | 2 (2) | 3 (8) | 2 (3) | 6 (17) | 2 (5) | 0 (0) | 2 (5) | 4 (8) | 3 (9)
Bundle branch block left (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cardiac flutter (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Asthenopia (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cataract (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Eye irritation (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Lacrimation increased (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Vision blurred (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Visual impairment (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vitreous floaters (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 2 (3) | 2 (2) | 1 (1) | 2 (2) | 0 (0)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 1 (1)
Ascites (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 2 (2) | 1 (1) | 2 (2) | 2 (2) | 2 (3) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (3) | 6 (8) | 3 (5) | 4 (5) | 1 (1) | 1 (1) | 2 (3) | 2 (3) | 3 (5)
Retching (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 2 (2) | 2 (3) | 3 (4) | 3 (3) | 1 (1) | 2 (3) | 1 (1) | 0 (0)
Asthenia (General disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Catheter site phlebitis (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest discomfort (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Chest pain (General disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Chills (General disorders) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Fatigue (General disorders) | 3 (3) | 6 (8) | 5 (6) | 5 (6) | 2 (2) | 0 (0) | 1 (1) | 4 (4) | 4 (4)
Influenza like illness (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Infusion site reaction (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mucosal inflammation (General disorders) | 1 (1) | 0 (0) | 2 (2) | 2 (2) | 1 (2) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Nodule (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 3 (4) | 3 (6) | 2 (2) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 2 (3)
Drug hypersensitivity (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypersensitivity (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lung infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Streptococcal bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (4) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Incision site pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (5) | 0 (0)
Scratch (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Antineutrophil cytoplasmic antibody increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood culture positive (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood glucose increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood magnesium decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Blood urine present (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Electrocardiogram qt prolonged (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Glomerular filtration rate decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haematocrit decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haemoglobin decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Weight decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
White blood cell count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (4)
White blood cell count increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 3 (3) | 2 (2) | 4 (4) | 2 (3) | 1 (1) | 1 (1) | 3 (3) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 4 (6) | 1 (1) | 3 (4) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperphosphatasaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (3) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Burning sensation (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 2 (2) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypogeusia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Paraesthesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Agitation (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Confusional state (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dysuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal pain (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vulvovaginal pruritus (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3) | 2 (2) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (4) | 2 (2) | 4 (7) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 2 (2)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasal mucosal discolouration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Paranasal sinus hypersecretion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rhinalgia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Hypoaesthesia facial (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Night sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (2) | 4 (4) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash pruritic (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin disorder (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Frontal sinus operation (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Flushing (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days